CLINICAL TRIAL: NCT02929849
Title: Influence of Herb With Alpha-glucosidase Properties (Salacia Chinensis) on Appetite, Glucose and Hormonal Factors: A Double Blind Randomized Placebo Controlled-crossover Trial
Brief Title: Satiety and Glucose Indices in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers University (Other)
Collaborators: OmniActive Health Technologies (Industry)
Responsible Party: Principal Investigator, Sue A. Shapses, Ph.D., RD, Professor, Rutgers University
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 10420
Record Dates: First submitted 2016-08-16; First posted 2016-10-11 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 300mg SC (Experimental): 300 mg Salacia Chinensis (SC). This will be compared to placebo.
  Interventions: Dietary Supplement: 300 mg SC
- 500mg SC (Active Comparator): 500 mg Salacia Chinensis (SC). This will be compared to placebo.
  Interventions: Dietary Supplement: 500 mg SC
- Placebo (Placebo Comparator): The investigators will examine subjects before and during a 3 hour period after subjects consume a Placebo capsule and a fixed breakfast meal.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 300 mg SC — Salacia (T1) capsule given with breakfast (mixed meal tolerance test)
  Arms: 300mg SC
Dietary Supplement: 500 mg SC — Salacia (T2) capsule given with breakfast (mixed meal tolerance test)
  Arms: 500mg SC
Dietary Supplement: Placebo — Placebo capsule given with breakfast (mixed meal tolerance test)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether an herb with known alpha-glucosidase inhibitor properties (Salacia Chinensis, SC), affects postprandial appetite ratings and glucose indices in overweight/obese individuals.

DETAILED DESCRIPTION:
Subjects are randomly assigned (double blinded) to 300 mg SC, 500 mg SC or placebo using a cross-over design on three different days (1 month wash out). Subjects consuming a capsule containing placebo or treatment(s) are examined before and after a fixed breakfast meal (50% carbohydrate; 30% fat; 20% protein).

Subjective appetite sensations are rated using visual analog scales (VAS) for hunger, satiety, fullness, and prospective food intake. In addition, the desire for specific tastes is analyzed and measurements are taken twice before breakfast (fasting baseline). After baseline screening and blood draw, postprandial appetite and taste perception ratings and blood will be obtained at multiple time points during the 3 hour postprandial period (30, 60, 90, 120,180 min). Blood will be analyzed for glucose/insulin, gut peptides, and other markers in response to the meal.

ELIGIBILITY:
Inclusion Criteria:

* BMI - overweight or stage 1 obesity
* Must be willing and able to visit the geographic vicinity of New Brunswick, NJ

Exclusion Criteria:

* (BP) [systolic BP> 140 and/or diastolic BP> 90]
* Fasting blood glucose >126
* Subject has a significant history or current presence of treated or untreated bleeding disorder, diabetes mellitus, thyroid disease, tachyarrhythmia, heart disease, kidney disease, or liver disease.
* History of chronic conditions and on prescription medication, surgery and or any treatment
* Any significant GI condition that would severely interfere with the evaluation of the study product including but not limited to inflammatory bowel disease (Ulcerative Colitis or Crohn's), history of frequent diarrhea, history of surgery for weight loss (including gastric bypass or lapband), history of perforation of the stomach or intestines, gastroparesis, clinically important lactose intolerance
* History or presence of all cancers in the prior two years.
* Participation in a clinical study with exposure to any registered and non-registered drug product within 30 days prior.
* Pregnant or lactating women.
* Subjects who are currently on any weight loss diets, weight loss regimen
* Subjects currently taking prescription medication for hypertension, cardiovascular disease, diabetes and/or other chronic conditions.
* Subject currently suffers from a sleep disorder and/or has a known history of (or is currently being treated for) clinical depression, eating disorder(s) or any other psychiatric condition(s), which in the opinion of the investigator, might put the subject at risk and/or confound the results of the study.
* Subject has a known allergy or sensitivity to any ingredient in the test product.
* Subject has any medical condition or uses any medication, nutritional product, dietary supplement or program, which in the opinion of the investigator, might interfere with the conduct of the study or place the subject at risk.
* Subject has a history of difficulty swallowing large pills or tablets.
* Investigator is uncertain about subject's capability or willingness to comply with the protocol requirements.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Appetite ratings (VAS) at either dose compared to placebo compared to placebo) | Change from Baseline and 3 hours
  Visual analog scale (VAS)

SECONDARY OUTCOMES:
Glucose indices (at either dose vs placebo) | Change from Baseline and 3 hours
  serum markers
Taste perception (dose compared to placebo) | Change from Baseline and 3 hours
  visual analog scale

OTHER OUTCOMES:
Appetite regulating hormones and other markers at either dose or placebo | Change from Baseline and 3 hours
  blood
Bone Turnover markers at either dose or placebo | Change from baseline over 3 hours
  blood

CONTACTS AND LOCATIONS:
Overall Officials: Sue Shapses, PhD, Principal Investigator — Rutgers University
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided
rules/regulations would need to be confirmed

REFERENCES:
- [Background] Kissileff HR, Thornton JC, Torres MI, Pavlovich K, Mayer LS, Kalari V, Leibel RL, Rosenbaum M. Leptin reverses declines in satiation in weight-reduced obese humans. Am J Clin Nutr. 2012 Feb;95(2):309-17. doi: 10.3945/ajcn.111.012385. Epub 2012 Jan 11. PMID 22237063
- [Background] Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. Int J Obes Relat Metab Disord. 2000 Jan;24(1):38-48. doi: 10.1038/sj.ijo.0801083. PMID 10702749
- [Background] Ibrugger S, Kristensen M, Mikkelsen MS, Astrup A. Flaxseed dietary fiber supplements for suppression of appetite and food intake. Appetite. 2012 Apr;58(2):490-5. doi: 10.1016/j.appet.2011.12.024. Epub 2012 Jan 5. PMID 22245724
- [Background] Hao L, Schlussel Y, Fieselmann K, Schneider SH, Shapses SA. Appetite and Gut Hormones Response to a Putative alpha-Glucosidase Inhibitor, Salacia Chinensis, in Overweight/Obese Adults: A Double Blind Randomized Controlled Trial. Nutrients. 2017 Aug 12;9(8):869. doi: 10.3390/nu9080869. PMID 28805670
- [Background] Kreitman A, Schneider SH, Hao L, Schlussel Y, Bello NT, Shapses SA. Reduced postprandial bone resorption and greater rise in GLP-1 in overweight and obese individuals after an alpha-glucosidase inhibitor: a double-blinded randomized crossover trial. Osteoporos Int. 2021 Jul;32(7):1379-1386. doi: 10.1007/s00198-020-05791-5. Epub 2021 Jan 11. PMID 33432459